CLINICAL TRIAL: NCT06781736
Title: Talking Circle for Native American Youth Living Well (AYoLi)
Brief Title: Talking Circle for Native American Youth
Acronym: AYoLi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00004266; 1UG3AT012547-01 (NIH)
Record Dates: First submitted 2025-01-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Mental Health Wellness 1; Behavior, Health; Emotional Stress
Keywords: mental well-being; emotional well-being; behavioral well-being
MeSH Terms: conditions — Health Behavior; Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Mental Health Wellness (mental, emotional and behavioral health issues)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mental Health Wellness 1 (Other): Talking Circle Intervention to promote the mental, emotional, and behavioral well-being
  Interventions: Behavioral: Talking Circle intervention

INTERVENTIONS:
Behavioral: Talking Circle intervention — Talking Circle intervention

SUMMARY:
Native American youth have higher rates of depression and lifetime major depressive episodes, and, by age 11, are more likely to have initiated alcohol and substance use than any other racial/ethnic group. The COVID19 pandemic only compounded this suffering--anxiety, stress, depression, substance use, and suicide related mental health disorders skyrocketed in many Native American communities, especially among youth. Though many are desperate for help, treatment options are scarce to non-existent. To meet this urgent need, our overarching objective is to leverage the empirically proven, highly effective, school based, Talking Circle intervention to promote the mental, emotional, and behavioral (MEB) health of geographically diverse (rural, urban) Native American youth. This study, "Talking Circle for Native American Youth Living Well (A Yo Li)" uses a Community Based Participatory Research (CBPR) approach to evaluate Talking Circle effectiveness, partnering with the United Keetoowah Band (UKB) of Cherokee Indians Tribe in Oklahoma, with members living in two geographically diverse areas, Adair County (rural), and Tulsa City (urban). "A Yo Li" in the UKB tribal language means "youth".

DETAILED DESCRIPTION:
Specific aims for Phase 1 (UG3) include:

UG3 Aim 1. To inform adaptation of the school-based Talking Circle intervention, a Community Partnership Committee (CPC) of UKB members will be developed to conduct a needs/asset mapping process to assess the needs, priorities, and resources for MEB health of UKB youth, paying special attention to the nuances of cultural difference between rural and urban UKB communities in Oklahoma.

UG3 Aim 2. To conduct a Talking Circle intervention Facilitator Training Program with rural and urban UKB tribal community members to catalyze capacity building and sustainability for future intervention.

UG3 Aim 3. To pilot the adapted evidenced-based Talking Circle intervention for the promotion of MEB health among (N=20) 10 to 12 year-olds UKB youth in Oklahoma.

ELIGIBILITY:
Inclusion Criteria:

* Native American students
* English speakers
* Read and write English
* At risk for mental health and behavioral health issues

Exclusion Criteria:

* Not Native American
* Non-English speakers
* Not able to read and write English
* Not at risk for mental health or behavioral health issues

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Native Reliance Questionnaire (NRQ) | Baseline and 3 month post-intervention
  24-items rated on a 5-point Likert scale to evaluate the presence of Native Reliance cultural identity; (minimum score of 24; maximum score of 120); higher score indicates a better outcome
Global Assessment of Individual Needs-Quick (GAIN-Q) | Baseline and 3 month post-intervention
  Subscales: Anxiety (7-items), ( minimum score of 0; maximum score of 7; lower score indicates better outcome) Stress (20-items; minimum score of 0; maximum score of 20; lower score indiciates better outcome) and Substance Use (16-items; minimum score of 0; maximum score of 16; lower score indicates better outcome)
Commercial Tobacco Use | baseline and 3 month post-intervention
  Global Youth Tobacco Survey (GYTS) a 43 item measure to assess key tobacco-control indicators, minimum score of 0; maximum score of 43 including use, cessation, and availability; lower score indicates better outcome

SECONDARY OUTCOMES:
Depression | baseline and 3 month post-intervention
  Center for Epidemiologic Studies Depression Scale Revised (CESD-R-10) a 10 item measure of depressed affect used in samples of NA youth with good reliability and validity (minimum score of 6; maximum score of 24) higher score is a worse outcome and lower score is a better outcome
Suicide Ideation | baseline and 3 month post-intervention
  Suicidal Ideation Questionnaire-Junior (SIQ-JR-15),15-items is rated on a 7-point scale indicating the frequency of suicidal thoughts, showing excellent validity and reliability, and an effective predictor of suicide risks in the Native American adolescent population (minimum score of 15 maximum score 105); the higher score indicates the greater risk of suicidal Ideation and lower score indicates lower risk of suicidal ideation.

CONTACTS AND LOCATIONS:
Locations (1):
- United Keetoowah Band of Cherokee Indians in Oklahoma, Tahlequah, Oklahoma, United States